CLINICAL TRIAL: NCT07184034
Title: Assessment of the Correlation Between Lipoprotein (a) Levels and Coronary Artery Findings on Multislice Computed Tomography
Brief Title: Lipoprotein a Assessment and Relation to Ca Score in CAD Patients Using MSCT
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Ayman Sobhy Kamel, Doctor, Assiut University
Other Study IDs: Lipoprotein a assessment
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate whether serum Lipoprotein(a) [Lp(a)] levels are associated with coronary artery calcium (CAC) score measured by multi-slice computed tomography (MSCT) in adults undergoing cardiac risk assessment.

The main questions it aims to answer are:

* Is there a correlation between elevated Lp(a) levels and higher CAC scores?
* Does Lp(a) provide additional predictive value for subclinical atherosclerosis beyond traditional cardiovascular risk factors?

Participants will:

* Undergo a non-contrast MSCT scan to measure CAC score.
* Provide a blood sample for measurement of Lp(a) and routine lipid profile.
* Have baseline clinical and demographic data collected, including cardiovascular risk factors.

DETAILED DESCRIPTION:
Lipoprotein(a) [Lp(a)] is a genetically determined lipoprotein particle structurally similar to LDL, with an additional apolipoprotein(a) component. Elevated Lp(a) levels have been identified as an independent and causal risk factor for atherosclerotic cardiovascular disease (ASCVD). The pro-atherogenic, pro-thrombotic, and pro-inflammatory properties of Lp(a) contribute to plaque development and vascular calcification.

Coronary artery calcium (CAC) score, assessed by non-contrast multi-slice computed tomography (MSCT), is a widely validated imaging biomarker of subclinical coronary atherosclerosis. CAC burden strongly predicts future cardiovascular events and is frequently used for individualized risk stratification. Recent studies suggest that individuals with elevated Lp(a) may also demonstrate higher CAC scores and faster progression of coronary calcification. However, the strength and consistency of this association remain insufficiently defined across different populations.

This observational study is designed to evaluate the correlation between serum Lp(a) levels and CAC score in adult participants undergoing cardiovascular risk assessment. Participants will undergo non-contrast MSCT scanning for CAC scoring, fasting blood sampling for Lp(a) and routine lipid profile, and collection of baseline demographic and clinical risk factors. Multivariable analyses will assess the independent relationship between Lp(a) and CAC score, as well as the potential incremental predictive value of Lp(a) beyond traditional risk factors such as LDL-C, hypertension, diabetes, and smoking.

We hypothesize that higher Lp(a) levels will be associated with higher CAC scores, independent of conventional cardiovascular risk factors, and that patients with both elevated Lp(a) and high CAC (≥100) will represent the subgroup at greatest risk for ASCVD. Demonstrating this relationship may improve cardiovascular risk stratification and highlight the importance of integrating Lp(a) measurement with imaging-based assessment in the early prevention of ASCVD.

ELIGIBILITY:
Inclusion Criteria:

* 1-adults aged 40-70

  * 2- classified as intermediate cardiovascular risk (10-20% 10 years ASCVD risk)
  * 3-undergoing MsCT for suspected coronary artery disease
  * 4- ability to provide informed consent

Exclusion Criteria:

* 1- known CAD or prior revascularization

  * 2-history of myocardial infarction or stroke
  * 3- statin or PCK9 inhibitor use in the past 3 months
  * 4-renal insufficiency (eGFR < 45ml/min/1.73m2)
  * 5-active inflammation or autoimmune disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult men and women aged 40 to 70 years who are classified as having intermediate cardiovascular risk (10-20% estimated 10-year ASCVD risk). Participants will be those referred for non-contrast multi-slice CT (MSCT) for suspected coronary artery disease and who are able to provide informed consent.
  Patients will be excluded if they have known coronary artery disease, prior myocardial infarction, prior coronary revascularization, or history of stroke. Additional exclusions include recent use of statins or PCSK9 inhibitors within the past 3 months, renal insufficiency (eGFR <45 mL/min/1.73m²), or active inflammatory or autoimmune disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between serum lipoprotein (a) levels and coronary artery calcium (CAC) score as measured by MSCT. | Baseline

SECONDARY OUTCOMES:
Check which of these patients will need revascularization after 6 to 12 months | Baseline

REFERENCES:
- [Background] Zeitouni M, Nanna MG, Sun JL, Chiswell K, Peterson ED, Navar AM. Performance of Guideline Recommendations for Prevention of Myocardial Infarction in Young Adults. J Am Coll Cardiol. 2020 Aug 11;76(6):653-664. doi: 10.1016/j.jacc.2020.06.030. PMID 32762899
- [Background] Kobayashi R, Kawakatsu S, Morioka D, Suzuki A. Diversity of dopamine transporter images in frontotemporal lobar degeneration-motor neuron disease. Psychogeriatrics. 2022 Sep;22(5):771. doi: 10.1111/psyg.12860. Epub 2022 Jun 5. No abstract available. PMID 35665572
- [Background] Thanassoulis G, Campbell CY, Owens DS, Smith JG, Smith AV, Peloso GM, Kerr KF, Pechlivanis S, Budoff MJ, Harris TB, Malhotra R, O'Brien KD, Kamstrup PR, Nordestgaard BG, Tybjaerg-Hansen A, Allison MA, Aspelund T, Criqui MH, Heckbert SR, Hwang SJ, Liu Y, Sjogren M, van der Pals J, Kalsch H, Muhleisen TW, Nothen MM, Cupples LA, Caslake M, Di Angelantonio E, Danesh J, Rotter JI, Sigurdsson S, Wong Q, Erbel R, Kathiresan S, Melander O, Gudnason V, O'Donnell CJ, Post WS; CHARGE Extracoronary Calcium Working Group. Genetic associations with valvular calcification and aortic stenosis. N Engl J Med. 2013 Feb 7;368(6):503-12. doi: 10.1056/NEJMoa1109034. PMID 23388002
- [Background] Hemmelgarn BR, Manns BJ, Lloyd A, James MT, Klarenbach S, Quinn RR, Wiebe N, Tonelli M; Alberta Kidney Disease Network. Relation between kidney function, proteinuria, and adverse outcomes. JAMA. 2010 Feb 3;303(5):423-9. doi: 10.1001/jama.2010.39. PMID 20124537
- [Background] Kamstrup PR, Benn M, Tybjaerg-Hansen A, Nordestgaard BG. Extreme lipoprotein(a) levels and risk of myocardial infarction in the general population: the Copenhagen City Heart Study. Circulation. 2008 Jan 15;117(2):176-84. doi: 10.1161/CIRCULATIONAHA.107.715698. Epub 2007 Dec 17. PMID 18086931
- [Background] Tsimikas S. A Test in Context: Lipoprotein(a): Diagnosis, Prognosis, Controversies, and Emerging Therapies. J Am Coll Cardiol. 2017 Feb 14;69(6):692-711. doi: 10.1016/j.jacc.2016.11.042. PMID 28183512
- [Background] Budoff MJ, Shaw LJ, Liu ST, Weinstein SR, Mosler TP, Tseng PH, Flores FR, Callister TQ, Raggi P, Berman DS. Long-term prognosis associated with coronary calcification: observations from a registry of 25,253 patients. J Am Coll Cardiol. 2007 May 8;49(18):1860-70. doi: 10.1016/j.jacc.2006.10.079. Epub 2007 Apr 20. PMID 17481445
- [Background] Greenland P, Blaha MJ, Budoff MJ, Erbel R, Watson KE. Coronary Calcium Score and Cardiovascular Risk. J Am Coll Cardiol. 2018 Jul 24;72(4):434-447. doi: 10.1016/j.jacc.2018.05.027. PMID 30025580